CLINICAL TRIAL: NCT01057355
Title: Endoscopic Ethanol Ablation of Communicating Pancreatic Cystic Neoplasms
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: slow accural
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark Topazian, Professor of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 009-004705; NCT01100229 (obsolete NCT alias)
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Neoplasms, Cystic, Mucinous, and Serous; Pancreatic Neoplasms; Ultrasonography, Interventional
Keywords: Intraductal papillary mucinous neoplasm; Mucinous cystic neoplasm; Endoscopic ultrasound; Endoscopic retrograde cholangiopancreatography; Pancreatic cyst; Pancreas cyst; Alcohol
MeSH Terms: conditions — Neoplasms, Cystic, Mucinous, and Serous; Pancreatic Neoplasms; Pancreatic Cyst | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cyst ethanol lavage (Experimental): Subjects receiving the study intervention
  Interventions: Procedure: EUS and/or ERCP with ethanol injections of pancreatic cyst

INTERVENTIONS:
Procedure: EUS and/or ERCP with ethanol injections of pancreatic cyst — Lavage of cyst with 80% ethanol
  Other Names: Alcohol lavage; Alcohol injection; Ethanol lavage; Ethanol injection; Endoscopic treatment; Pancreas cyst ablation

SUMMARY:
Pancreatic cysts are common, and some pancreas cysts have malignant potential. Usual treatment of these cysts is either observation or surgical removal of part or all of the pancreas. Minimally invasive treatment via endoscopy has been described, using endoscopic ultrasound (EUS) guided ethanol injections. Such studies exclude cysts that communicate with the main pancreatic duct, to avoid burning the main pancreatic duct with ethanol. In this study, pancreas cysts communicating with the main pancreas duct are treated with ethanol via endoscopic retrograde cholangiopancreatography (ERCP) and/or EUS.

DETAILED DESCRIPTION:
Subjects will undergo EUS and/or ERCP as outpatients. For cysts shown to communicate with the main pancreas duct, a balloon catheter will be placed in the main pancreatic duct via ERCP. The balloon catheter will isolate the cyst from the main pancreatic duct, allowing ethanol injections of the cyst. A pancreatic duct stent will be placed in some patients, requiring repeat endoscopy for removal at another time.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a pancreatic cystic lesion, at least 2 cm in maximum diameter
* Cyst may communicate, or definitely communicates, with the pancreatic duct (based on prior CT, MR, ERCP, or EUS images)
* Treatment of the cystic lesion is desired due to symptoms or concern for subsequent malignancy
* Age at least 18 years
* Able to give informed consent
* Surgical treatment has been considered and a surgical consultation offered to the patient, OR the subject's cyst does not meet consensus criteria for surgical resection. (Current consensus criteria for resection are one or more of the following: cyst is symptomatic, ≥ 3 cm in diameter, contains a mural nodule, cytology of cyst fluid is positive for malignancy, or main pancreatic duct diameter is > 6 mm.)

Exclusion Criteria:

* Known or suspected pregnancy, or nursing
* History of pancreatitis within 3 months prior to study endoscopy procedures
* Cyst has a primarily microcystic architecture on EUS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events requiring treatment or hospitalization | 3 days, 30 days
Decrease in volume of the pancreatic cyst by cross-sectional imaging studies (CT or MR) performed before and after treatment | 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Topazian, M.D., Principal Investigator — Mayo Clinic